CLINICAL TRIAL: NCT04759950
Title: Effects of Combined Therapies of Physical Exercise, Mindfulness and Cognitive Stimulation on Cognition and Neuroplasticity in Chronic Stroke Patients: A Randomized Controlled Trial
Brief Title: Exercise the Mind and Brain. A Multimodal Intervention in Stroke
Acronym: Mindfit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Collaborators: Fundació La Marató de TV3 (Other); Germans Trias i Pujol Hospital (Other); Institut Guttmann (Other); Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other); University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Maria Mataro Serrat, Professor, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: University of Barcelona; 201717.30.31.32 (Other Grant/Funding Number: La Marato de TV3)
Record Dates: First submitted 2020-12-31; First posted 2021-02-18 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Stroke
Keywords: Neuroplasticity; stroke; neuroprotection; physical exercise; cognitive training; mindfulness; neuroimaging; intervention; randomization; blind
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Intervention Model Description: 141 participants at 3 to 60 months after stroke are randomly allocated to one of three arms: The first group (n=47) receives computer-based cognitive training (CCT) combined with a multicomponent physical exercise program. The second group (n=47) receives CCT combined with mindfulness-based stress reduction therapy. Finally, the third group (n=47), as an active control group, receives only CCT.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The randomization sequence is concealed (blinded) from research personnel, so that the investigators are not aware of whether a particular subject has been randomized to one of the intervention groups or to the active control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Physical exercise & cognitive training group (Experimental): The Physical exercise & cognitive training group receives a multicomponent physical exercise program combined with computer-based cognitive training.
  Interventions: Behavioral: Multicomponent Physical Activity Program; Behavioral: Computerized Cognitive Training
- Mindfulness & cognitive training group (Experimental): The Mindfulness & cognitive training group receives mindfulness-based stress reduction therapy combined with computer-based cognitive training.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction Program; Behavioral: Computerized Cognitive Training
- Cognitive training group (Active Comparator): The Cognitive training group, as an active control group, receives only computer-based cognitive training.
  Interventions: Behavioral: Computerized Cognitive Training

INTERVENTIONS:
Behavioral: Multicomponent Physical Activity Program — The proposed physical exercise intervention follows the American College of Sports Medicine (ACSM, 2017) and the American Stroke Association (Billinger et al., 2014) recommendations for stroke patients. The five weekly 45-minute sessions are divided into (1) three sessions guided and supervised telematically by a physical exercise specialist and a physiotherapist; (2) and two autonomous exercise sessions. The supervised sessions include exercises to work aerobic capacity, muscle strength and endurance, flexibility, agility, and balance. The intensity of these exercises is prescribed individually according to each participant's initial level and are gradually increased as the program progresses. Participants are encouraged to walk at a similar intensity on autonomous physical exercise days as performed in the guided sessions (moderate intensity), based on the Borg scale of perceived exertion (Borg, 1982).
  Arms: Physical exercise & cognitive training group
Behavioral: Mindfulness-Based Stress Reduction Program — This intervention follows an adaptation of the scheme and instructions of the official Mindfulness-Based Stress Reduction (MBSR) program designed by Jon Kabat-Zinn. It includes body scanning, sitting meditation, and gentle hatha yoga techniques. An accredited mindfulness instructor leads the 12-week online program, which comprises a presentation session, followed by eight intervention sessions (once a week, lasting 2.5 hours) and an intensive practice session interspersed between sessions six and seven. Apart from the supervised session, the therapist asks participants to carry out some independent practice daily.
  Arms: Mindfulness & cognitive training group
Behavioral: Computerized Cognitive Training — An accredited neuropsychologist programs and supervises the computerized cognitive training through the Guttmann Neuropersonal Trainer (GNPT®) platform. The 12-week program consists of five sessions a week (45 minutes each) that include personalized activities planned to stimulate executive functioning, attention, processing speed, and memory.

SUMMARY:
The main objective of MindFit Project is to develop an evidence-based multimodal investigation of combined non-pharmacological strategies in chronic stroke patients and clarify the neuroplasticity mechanisms underlying the benefits of physical exercise and mindfulness strategies combined with cognitive training on post-stroke recovery. The investigators have adopted a multidisciplinary and multimodal approach to provide a more integrative perspective using cognitive, social-psychological, biochemical, and neuroimaging measurements.

DETAILED DESCRIPTION:
The MindFit Project is a multicentric, prospective, parallel, single-blinded, randomized controlled trial with a sample of 141 participants at 3 to 60 months after stroke. Participants are randomly allocated to one of three arms (through a simple randomizing procedure with a 1:1:1 ratio created with a random sequence generator software).

The first group (n=47) receives computer-based cognitive training (CCT) combined with a multicomponent physical exercise program. The second group (n=47) receives CCT combined with mindfulness-based stress reduction therapy. Finally, the third group (n=47), as an active control group, receives only CCT. All interventions last 12 weeks.

Within two weeks before the start of the interventions, and again at 3 months after completing the interventions, medical, cognitive, and physical assessments, neuroimaging, and biological samples collection are performed.

The objectives of this project are:

1. To examine the effects of multimodal interventions in a population of chronic stroke patients on various domains: cognition, emotion, physical health, and quality of life.
2. To examine specific plasticity effects of each of the three interventions regarding structural and functional magnetic resonance imaging (MRI) and how these changes may contribute to cognitive and emotional benefits.
3. To study the molecular mechanisms by which the different types of interventions influence cognitive, emotional and brain benefits.
4. To study interventions-induced microbiome changes and to explain how these changes may induce inflammatory and immune responses that may contribute to cognitive, emotional and brain benefits.
5. To determine the demographic, clinical and genetic factors that may modulate cognitive, emotional and brain changes: baseline cognitive status; baseline cerebral status (atrophy, total intracranial volume); sex; age, educational level, intelligence.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-80 years old
* Ischemic or hemorrhagic stroke
* Stroke diagnoses between 3-60 months ago
* To have consent from a physician to engage in an exercise intervention
* Fluency in Catalan or Spanish (I.e., able to understand and speak)
* Accept to take part in the study and sign the informed consent according to the Declaration of Helsinki.

Exclusion Criteria:

* Cognitive impairment (MMSE > 23)
* Severe aphasia (item 9 of the NIHSS scale ≥ 2)
* Severe sensory problems
* Other neurological conditions apart from stroke
* Severe pre-stroke psychiatric disorders (e.g., bipolar disorder, schizophrenia)
* History of alcohol or other toxic abuse

Exclusion criteria only for MRI examination:

* Claustrophobia
* Medical device (e.g., pacemaker implants, stents)
* Other metal objects in the body

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Change in immediate verbal attention after receiving treatment | 3 months (at baseline, 3 months from baseline)
  Forward Digit Span (WAIS III)
Change in verbal digit working memory after receiving treatment | 3 months (at baseline, 3 months from baseline)
  Backward Digit Span (WAIS III)
Change in verbal memory after receiving treatment | 3 months (at baseline, 3 months from baseline)
  Rey Auditory Learning Test
Change in visual memory after receiving treatment | 3 months (at baseline, 3 months from baseline)
  Rey's Complex Figure Test
Change in executive function, verbal fluency after receiving treatment | 3 months (at baseline, 3 months from baseline)
  Phonetic Fluency is measured using the Controlled Oral Word Association Test, spanish adaptation, and semantic fluency test using the category Animal
Change in executive function, inhibition after receiving treatment | 3 months (at baseline, 3 months from baseline)
  Stroop Test
Change in executive function, set-switching task after receiving treatment | 3 months (at baseline, 3 months from baseline)
  Trail Making Test
Change in language, naming after receiving treatment | 3 months (at baseline, 3 months from baseline)
  Boston naming Test

SECONDARY OUTCOMES:
Changes in psychological distress | 3 months (at baseline, 3 months from baseline)
  Clinical Outcomes in Routine Evaluation (CORE-OM)
Changes in depression and anxiety | 3 months (at baseline, 3 months from baseline)
  Depression Anxiety Stress Scale (DASS-21)
Changes in wellbeing | 3 months (at baseline, 3 months from baseline)
  Ryff Scales of Psychological Wellbeing.
Changes in Mindfulness | 3 months (at baseline, 3 months from baseline)
  Mindful Attention Awareness Scale (MAAS)
Changes in White matter integrity | 3 months (at baseline, 3 months from baseline)
  White matter integrity: tractography
Changes in Resting-state connectivity | 3 months (at baseline, 3 months from baseline)
  Resting state brain activity using fMRI
Changes in brain volumetry | 3 months (at baseline, 3 months from baseline)
  Grey and white matter volume measured by MRI
Molecular changes: growth factors (BDNF, SDF1-a, VEGF-A, IGF-1, and NGF), cortisol, protein C reactive, IL-6 and homocysteine levels | 3 months (at baseline, 3 months from baseline)
  Quantification of different biomarkers from blood samples.
Changes in Microbiota data | 3 months (at baseline, 3 months from baseline)
  Bacterial composition of stool samples in terms of relative abundance
Changes in Sleep | 3 months (at baseline, 3 months from baseline)
  Pittsburgh Sleep Quality Index (PSQI)
Changes in Fitness | 3 months (at baseline, 3 months from baseline)
  Senior Fitness Test (SFT)
Changes in stroke specific quality of life | 3 months (at baseline, 3 months from baseline)
  Stroke-specific Quality of Life Scale (ECVI-38)
Changes in quality of life | 3 months (at baseline, 3 months from baseline)
  World Health Organization Quality of Life (WHOQOL-BREF)
Changes in mental fatigue | 3 months (at baseline, 3 months from baseline)
  Fatigue Assessment Scale (FAS)
Changes in physical activity: | 3 months (at baseline, 3 months from baseline)
  Spanish version of the reduced Minnesota leisure-time physical and activity questionnaire (VREM)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Mataro, PhD, Principal Investigator — University of Barcelona
Locations (1):
- Maria Mataro, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bermudo-Gallaguet A, Ariza M, Agudelo D, Camins-Vila N, Boldo M, Ferrer-Uris B, Busquets A, Pera G, Caceres C, Gomis M, Dacosta-Aguayo R, Clemente IC, Garcia-Molina A, Mata MJD, Toran-Monserrat P, Erickson KI, Mataro M. Effects of mindfulness and exercise on cognition and emotion in adults with mild deficits in the chronic post-stroke phase: A randomized controlled trial. Ann Phys Rehabil Med. 2025 Oct;68(7):102008. doi: 10.1016/j.rehab.2025.102008. Epub 2025 Aug 21. PMID 40845631
- [Derived] Bermudo-Gallaguet A, Ariza M, Dacosta-Aguayo R, Agudelo D, Camins-Vila N, Boldo M, Carrera O, Vidal S, Ferrer-Uris B, Busquets A, Via M, Pera G, Caceres C, Gomis M, Garcia-Molina A, Tormos JM, Arrabe A, Diez G, Dura Mata MJ, Toran-Monserrat P, Soriano-Raya JJ, Domenech S, Perera-Lluna A, Erickson KI, Mataro M. Effects and mechanisms of mindfulness training and physical exercise on cognition, emotional wellbeing, and brain outcomes in chronic stroke patients: Study protocol of the MindFit project randomized controlled trial. Front Aging Neurosci. 2022 Sep 29;14:936077. doi: 10.3389/fnagi.2022.936077. eCollection 2022. PMID 36248000